CLINICAL TRIAL: NCT00937469
Title: Social Skills Training and Standard Treatment Versus Standard Treatment of Children With ADHD - Attention Deficit Hyperactivity Disorder. Attachment Problems Among Children With ADHD
Brief Title: Social Skills Training and Standard Treatment Versus Standard Treatment of Children With Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: SOSTRA-ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Zealand (Other)
Collaborators: Zealand University Hospital (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Region Sjælland (Other)
Responsible Party: Ole Jakob Storebø, Psychologist. MS, Børne- og Ungdomspsykiatrisk Afdeling, Region Sjælland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOSTRA-BU/REGIONSJ.1; Ethics C. no. SJ-85; Data p. agency no. DO50892
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-07

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder
Keywords: Social skills training for children with ADHD; Children with ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Behavior Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Social sk. tr., parent tr.,standard tr. (Experimental)
  Interventions: Behavioral: Social skills training, parental tr. and standard tr.
- Standard treatment (Active Comparator)
  Interventions: Other: Standard treatment

INTERVENTIONS:
Behavioral: Social skills training, parental tr. and standard tr. — Social skills training will consist of 8 weeks of group treatment with weekly sessions of one and a half hours and includes role play, exercises and games as well as home work which will include the parents. At the same time the parents are participating in parental training groups,that will focus on supporting the children's social training. Both the children and the parental groups are lead by two group therapists. The intervention will be additional to the received standard treatment.
  Other Names: Psychosocial treatment.; Behavioral treatment.
  Arms: Social sk. tr., parent tr.,standard tr.
Other: Standard treatment — The standard treatment consists of medical treatment, briefing, consulting and supporting conversations with a focus on securing compliance to the treatments´ and on aiding children and their families with the difficulties arising with the children's illness. Furthermore the parents participate in parental groups three times during the 8 weeks in which the experiment takes place. This group lasts 2 hours and is managed by two nurses who are attached to the ADHD- treatment group.
  Other Names: Treatment as usual.
  Arms: Standard treatment

SUMMARY:
The primary purpose of the trial is to examine the effect of the combination of social skills training, parental training and standard treatment versus standard treatment in ADHD patients.

The secondary purpose is to examine differences in the effect of the treatment in relation to the different competences of attachment: secure attachment: unsecure dismissing, unsecure preoccupied or disorganized attachment and in the categories; emotional openness, balance of positivity / negativity to attachment figure/s, idealisation of attachment figure/s, dismissal and/or derogation of attachment, the ability of conflict resolution, disorganisation and coherence of the narrative description.

The tertiary purpose of the trial is to examine differences in the effect of the treatment in relation to the degree of parents symptoms of ADHD.

DETAILED DESCRIPTION:
Background:

Many children with ADHD have, beside the main symptoms hyperactivity, impulsivity and a lack of ability to maintain attention, difficulties with social interaction. This is a burden in the childrens relationship towards parents, peers and teachers and thereby influencing their performances in school. Many children with ADHD find great help in receiving medical treatment, which has a good effect on the children's problems with hyperactivity, impulsivity and lacking attention. However, social interaction problems will probably not be set right due to medication alone. Several studies have shown that social skills training can help children with ADHD in their social interactions. It is also an interesting issue to further investigate treatment effect in relation to the ADHD-children's attachment competences, as one must assume that differences in attachment competences may influence the children's relationship and social interaction problems.

The research intervention:

Social skills training will consist of 8 weeks of group treatment with weekly sessions of one and a half hours and includes role play, exercises and games as well as home work which will include the parents. At the same time the parents are participating in parental training groups,that will focus on supporting the children's social training. Both the children and the parental groups are lead by two group therapists. The intervention will be additional to the received standard treatment.

Control treatment:

The standard treatment consists of medical treatment, briefing, consulting and supporting conversations with a focus on securing compliance to the treatments´ and on aiding children and their families with the difficulties arising with the children's illness. Furthermore the parents participate in parental groups three times during the 8 weeks in which the experiment takes place. This group lasts 2 hours and is managed by two nurses who are attached to the ADHD- treatment group.

Method:

Children in the age of 8-12 years with a diagnosis of ADHD are randomised to either the combination standard treatment, social skills training with parental training or to standard treatment. The sample size calculation shows that 52 patients must be included in the trial to show a 4 point difference in the primary outcome. The examinations of the children will take place at the baseline and after three and six months.

Experimental hypotheses

1. There is significant difference between the clinical effect of the combination social skills training, parental training and standard treatment versus standard treatment 3 and 6 months after the beginning of the treatment in relation to the children's social competences.

   Measures: sub index 'Social Problems' from Conners CBRS and the sub index 'Peer Relations' from Conners 3.
2. There is significant difference between the clinical effect of the combination social skills training, parental training and standard treatment versus standard treatment 3 and 6 months after the beginning of the treatment in relation to hyperactivity/impulsivity problems.

   Measured by: sub index 'Hyperactivity/Impulsivity' from Conners 3.
3. There is significant difference between the clinical effect of the combination social skills training, parental training and standard treatment versus standard treatment 3 and 6 months after the beginning of the treatment in relation to the amount of children's aggressive behaviour and the children's emotional distress.

   Measures: sub indexes from Conners CBRS: 'Aggressive Behaviour' and 'Emotional distress'.
4. There is significant difference between the clinical effect of the combination social skills training, parental training and standard treatment versus standard treatment 3 and 6 months after the beginning of the treatment in relation to the childrens academic performance and executive functioning.

   Measures: sub indexes 'Academic Difficulties' from Conners CBRS and 'Executive Functioning' from Conners 3.
5. There is significant difference between the clinical effect of the combination social skills training, parental training and standard treatment versus standard treatment 3 and 6 months after the beginning of the treatment in relation to the children's social competences and symptoms of ADHD in relation to the different competences of attachment.

   Measured by: CAI- Children Attachment Interview.
6. There is significant difference between experimental and standard treatment 6 months after start of treatment, as reflected in positive changes in the childrens attachment skills or an improvement in the categories; emotional openness, balance of positivity / negativity to attachment figure/s, idealisation of attachment figure/s, dismissal and/or derogation of attachment, the ability of conflict resolution, disorganisation and coherence of the narrative description.

   Measured by: CAI- Children Attachment Interview
7. There is significant difference between the clinical effect of the combination social skills training, parental training and standard treatment versus standard treatment 3 and 6 months after the beginning of the treatment in relation to the children's social competences and symptoms of ADHD in relation to the parent's amount of ADHD symptoms.

Measured by: ASRS Symptom Checklist.

Null hypothesis

* There is no significant difference between the clinical effect of the combination social skills training, parental training and standard treatment versus standard treatment 3 and 6 months after the beginning of the treatment.
* There is no difference in the effect in one or the other treatment if the children's different forms of attachment styles are considered
* There is no difference in the effect in one or the other treatment if the children's parents ADHD symptoms are considered There is no difference 6 month after the beginning of the treatment in the effect in one or the other treatment if the childrens attachment skills or the undercategories are considered 6 month after the beginning of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The parents should be interested in taking part in parental groups in Børnepsykiatrisk Ambulatorium in Holbæk.
2. The patients (and the parents) must understand and speak Danish language to an extent where a translator is not needed in order to be able to complete the assessment and the treatment.
3. The patients´ parents must give informed consent to participate in the trial.
4. The children must be between 8-12 years old by the time of the start of the assessment.
5. Both boys and girls can participate.
6. Children with a total verbal or nonverbal IQ>80 according to the WISC III.
7. The children must fulfil research criteria for the diagnosis ADHD according to DSM IV (1994): 314.00, 314.01,314.02 or 314.9.
8. The parents must be prepared to the fact that their children have to receive medical treatment for their ADHD.

Exclusion Criteria:

Patients with the following diagnoses according to DSM IV:

1. Schizophrenia:

   295.30(Paranoid type) 295.10(Disorganized type) 295.20(Catatonic type) 295.90(Undifferentiated type) 295.60(Residual type) 295.70(Schizoaffective Disorder) 297.1(Delusional Disorder) 298.8(Brief Psychotic Disorder) 297.3(Shared Psychotic Disorder) 298.9(Psychotic Disorder Not Otherwise Specified)
2. Children with autism according to DSM IV:

   299.00 (Autistic Disorder) 299.10 (Childhood Disintegrative Disorder) 299.80 (Asperger´s Disorder) or a cut of score on both the SCQ questionnaires >15.
3. Violent and criminal youngsters.
4. Children with a total verbal or nonverbal IQ<80 according to WISC III
5. Strong resistance from the child against participating.
6. Previous started medical treatment for ADHD.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
ADHD core symptoms: measured by Conners 3 index: 'Hyperactivity- Impulsivity Scale' (teacher rated.) | 3 month
ADHD core symptoms: measured by Conners 3 index: 'Hyperactivity- Impulsivity Scale' (teacher rated.) | 6 month

SECONDARY OUTCOMES:
Aggressive behaviour: measured by Conners CBRS; subscale: 'Aggressive Behaviour Scale' (teacher rated). | 3 months
Emotional distress: measured by Conners CBRS: subscale: 'Emotional Distress Scale' (teacher rated). | 3 months
Executiv functioning: measured by Conners 3 index: 'Executive Functioning' (teacher rated). | 3 month
Academic difficulties: measured by Conners CBRS index: 'Academic Difficulties' (teacher rated). | 3 month
Attachment: measured by Children Attachment Interview. | 6 month
Aggressive behaviour: measured by Conners CBRS; subscale: 'Aggressive Behaviour Scale' (teacher rated). | 6 month
Emotional distress: measured by Conners CBRS: subscale: 'Emotional Distress Scale' (teacher rated). | 6 month
Executiv functioning: measured by Conners 3 index: 'Executive Functioning' (teacher rated). | 6 month
Academic difficulties: measured by Conners CBRS index: 'Academic Difficulties' (teacher rated). | 6 month
Social Skills: measured by Conners CBRS subscale: 'Social Problems Scale'( teacher rated) and by Conners 3 subscale: 'Peer Relations Scale'. (teacher rated). | 3 month
Social Skills: measured by Conners CBRS subscale: 'Social Problems Scale'( teacher rated) and by Conners 3 subscale: 'Peer Relations Scale'. (teacher rated). | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Pedersen, MD,Phd., Study Director — Region Sjælland
Locations (1):
- Børnepsykiatrisk Ambulatorium, Børne- og Ungdomspsykiatrisk Afdeling, Region Sjælland, Holbæk, Denmark

REFERENCES:
- [Derived] Storebo OJ, Gluud C, Winkel P, Simonsen E. Social-skills and parental training plus standard treatment versus standard treatment for children with ADHD--the randomised SOSTRA trial. PLoS One. 2012;7(6):e37280. doi: 10.1371/journal.pone.0037280. Epub 2012 Jun 20. PMID 22745657
- [Derived] Storebo OJ, Pedersen J, Skoog M, Thomsen PH, Winkel P, Gluud C, Simonsen E. Randomised social-skills training and parental training plus standard treatment versus standard treatment of children with attention deficit hyperactivity disorder - the SOSTRA trial protocol. Trials. 2011 Jan 21;12:18. doi: 10.1186/1745-6215-12-18. PMID 21255399
- See also: Related Info — http://regionsjaelland.dk